CLINICAL TRIAL: NCT02183233
Title: A Double-blind Randomized, Placebo Controlled Study to Assess the Efficacy and the Safety of Eschscholtzia Californica 1000 mg Per Day in Treating Primary Insomnia During a 28 Day Treatment Duration.
Brief Title: Efficacy and Safety of Eschscholtzia Californica in Treating Primary Insomnia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1120.2
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

ARMS (2):
- Eschscholtzia Californica (Experimental)
  Interventions: Drug: Eschscholtzia Californica
- Eschscholtzia Californica Placebo (Placebo Comparator)
  Interventions: Drug: Eschscholtzia Californica Placebo

INTERVENTIONS:
Drug: Eschscholtzia Californica
  Arms: Eschscholtzia Californica
Drug: Eschscholtzia Californica Placebo
  Arms: Eschscholtzia Californica Placebo

SUMMARY:
The aim of this trial was to assess the efficacy and safety of Eschscholtzia Californica (EC) in treating patients having psycho-physiologic insomnia in a double-blind randomised placebo controlled trial during a 28-day treatment duration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female above 18 or below 65 years old
* Diagnosis of psycho-physiologic insomnia, according to the criteria of DSM-IV (Diagnostic and Statistical manual - Version IV)
* Written informed consent

Exclusion Criteria:

* Patient who is already taking other investigational drugs or who has taken part in another trial during the past three months
* Patient who has an history of psychiatric diseases, such as:

  * anxiety disorders; the score of the HAMA (Hamilton anxiety scale) must be < 10
  * depression according to the DSM IV criteria; the score of the HAMD (Hamilton depression scale) must be < 10
  * mania
  * schizophrenia
  * dementia
* Patient who has an history of neurologic diseases, such as:

  * Parkinson syndrome
  * crania cerebral trauma post syndrome
  * brain tumor
  * fibromyalgia
* Patient who has an history of an iatrogenic insomnia, due to drugs like antidepressor, neuroleptic or benzodiazepine, hypnotic
* Patient with an hypersomnia or a sleep apnea syndrome
* Patient with any pathology inducing a chronic pain, a pyrosis, a nocturnal pollakiuria, a dyspnea
* Patient with a Restless Leg Syndrome
* Patient with severe hepatic or renal insufficiency which judged to be regarded as clinically relevant by the investigator, or any known clinically significant disease which may induce a risk for the patient in participating to the trial
* Breast feeding or pregnant female, or female with no efficient contraception method
* Patient with non-stabilised thyroid dysfunction
* Patient with a known allergy to Eschscholtzia Californica or its compounds
* Patient with alcohol or drug dependency
* Patient drinking tea, coffee or Coca-Cola after 4 p.m.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 1998-01; Primary Completion 1998-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sleep latency | Days 0, 7, 14 and 28

SECONDARY OUTCOMES:
Change from baseline in sleep duration | Days 0, 7, 14 and 28
Change from baseline in number of awakenings | Days 0, 7, 14 and 28
Change from baseline in quality of sleep | Days 0, 7, 14 and 28
Change from baseline in presence of morning sleepiness | Days 0, 7, 14 and 28
Change from baseline in morning concentration ability | Days 0, 7, 14 and 28
Change from baseline in Clinical Global Impression (CGI) score | Days 0, 7, 14 and 28
Change from baseline in quality of life (QL questionnaire SF-23) | Days 0, 7, 14 and 28
Number of patients with adverse events | up to 28 days